CLINICAL TRIAL: NCT02624154
Title: Pancreatic Neuroendocrine Tumor：Factor of Surgery Influencing Survival
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Qinchang Chen, Principal Investigator, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: SYSU 211
Record Dates: First submitted 2015-11-30; First posted 2015-12-08 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-11

CONDITIONS: Pancreatic Neuroendocrine Tumor
MeSH Terms: conditions — Adenoma, Islet Cell | interventions — Pancreatectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: pancreatectomy — Remove the pancreatic neuroendocrine tumor by surgery

SUMMARY:
Investigator determined the factor of surgery associated with the survival of pancreatic neuroendocrine tumor.

DETAILED DESCRIPTION:
The variables including clinical characteristics, surgical data and pathological findings are examined by univariate and multivariate analyses.

ELIGIBILITY:
Inclusion Criteria:

* The patients with pancreatic neuroendocrine tumor underwent pancreatectomy

Exclusion Criteria:

* The patients with pancreatic neuroendocrine tumor did not undergo pancreatectomy

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Investigators selected the patient who underwent pancreatectomy during the time from 2010 to 2013 at the First Affiliated Hospital of Sun Yat-sen University.
Sampling Method: Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The survival rate | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Shaowei Gao, Doctor, Study Director — First Affiliated Hospital, Sun Yat-Sen University